CLINICAL TRIAL: NCT02025985
Title: A Phase II, Open-label Study of Efficacy and Safety of the Selective Inhibitor of Nuclear Export/SINE™ Compound KPT-330 (Selinexor) in Patients With Advanced Gynaecologic Malignancies
Brief Title: Study of KPT-330 (Selinexor) in Female Patients With Advanced Gynaecologic Malignancies
Acronym: SIGN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-005; 2013-003650-24 (EudraCT Number)
Record Dates: First submitted 2013-12-27; First posted 2014-01-01 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Carcinoma; Endometrial Carcinoma; Cervical Carcinoma
Keywords: Karyopharm; KPT-330; Selinexor; SIGN; ovarian cancer; endometrial cancer; cervical cancer; SINE™; HER2 negative
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort A-Ovarian carcinoma: Selinexor up to 60 mg/m^2 BIW (Experimental): Participants with ovarian carcinoma who were platinum refractory or platinum resistant and had received at least one line of chemotherapy for relapsed disease received a dose of 50 milligram per meter square (mg/m^2) of selinexor oral tablets twice weekly (BIW) (doses at least 36 hours apart) with light meal and 120 milliliters (mL) of water in a 4-week treatment cycles. After 12 weeks of treatment, a dose of 60 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 once weekly (QW). This treatment continued until progression of disease (PD) or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
  Interventions: Drug: Selinexor
- Part 1: Cohort B-Endometrial carcinoma: Selinexor up to 60 mg/m^2 BIW (Experimental): Participants with endometrial carcinoma who had received at least one line of chemotherapy for relapsed or advanced (Stage IVb, IIIc) disease received a dose of 50 mg/m^2 of selinexor oral tablets BIW (doses at least 36 hours apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 12 weeks of treatment, a dose of 60 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
  Interventions: Drug: Selinexor
- Part 1: Cohort C-Cervical carcinoma: Selinexor up to 60 mg/m^2 BIW (Experimental): Participants with cervical carcinoma who had received at least one line of chemotherapy for relapsed or advanced (Stage IV) disease received a dose of 50 mg/m^2 of selinexor oral tablets BIW (doses at least 36 hours apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 12 weeks of treatment, a dose of 60 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
  Interventions: Drug: Selinexor
- Part 2: Cohort A-Ovarian carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW (Experimental): Participants with ovarian carcinoma who were platinum refractory or platinum resistant and had received at least one line of chemotherapy for relapsed disease received a dose of 35 mg/m^2 of selinexor oral tablets BIW (doses at least 36 hours apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 6 weeks of treatment, a dose of 50 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
  Interventions: Drug: Selinexor
- Part 2: Cohort A-Ovarian carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW (Experimental): Participants with ovarian carcinoma who were platinum refractory or platinum resistant and had received at least one line of chemotherapy for relapsed disease received a dose of 50 mg/m^2 of selinexor oral tablets QW (doses at least 5 days apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 6 weeks of treatment, a dose of 60 mg/m^2 of selinexor oral tablets QW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Route of administration and dosage form: Oral tablet; Doses: 35 mg/m^2 BIW, 35 mg/m^2 QW, 50 mg/m^2 BIW, 50 mg/m^2 QW, 60 mg/m^2 BIW, 60 mg/m^2 QW.
  Treatment cycles were 4 weeks each i.e., 28 day cycles.
  Other Names: KPT-330; XPOVIO

SUMMARY:
The primary trial objective is to determine the efficacy of KPT-330 (selinexor) in participants with advanced or metastatic gynaecological cancers by disease control rate (complete response (CR) or partial response (PR) or stable disease (SD) for at least 12 weeks, assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

DETAILED DESCRIPTION:
Two-stage Phase 2 study in 3 separate gynecological cancer cohorts, with an additional set of participants in the ovarian cohort randomized into 2 different treatment regimens. The study is divided between a Primary Treatment Phase and a Maintenance Phase with each phase supported by a separate database.

Part 1 - Three parallel cohorts of participants with ovarian (Cohort A), endometrial (Cohort B), or cervical (Cohort C) carcinoma were enrolled.

Part 2 - Based on the observed tolerability and efficacy profile in the ongoing ovarian cohort (Cohort A), 2 additional treatment schedules will be explored to optimize the dosing schedule in a participant population with ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate hematologic function defined as:

  * platelets ≥125*10^9 per liter (/L)
  * hemoglobin ≥5.59 millimoles per liter (mmol/L) or 9 grams per deciliter (g/dL)
  * Absolute neutrophil count (ANC) ≥1.5*10^9/L
  * White blood cells (WBC) count ≥3.0*10^9/L
  * Up to 5 percent (%) deviation is tolerated. Transfusions and growth factors are allowed.
* Adequate liver function defined as adequate hepatic function within 14 days prior to Cycle 1 Day 1: total bilirubin <2 times the upper limit of normal (ULN) (except participants with Gilbert's syndrome, who must have a total bilirubin of <3 times ULN), aspartate aminotransferase (AST) <2.0 times ULN, and alanine aminotransferase (ALT) <2.0 times ULN. In the case of known (radiologically and/or biopsy- documented) liver metastasis, AST <5.0 times ULN and ALT <5.0 times ULN is acceptable. Up to 10% deviation is acceptable.
* Renal function defined as a calculated or measured glomerular filtration rate ≥30 milliliter per minute (mL/min).
* The participant has recovered to Grade less than or equal to (≤) 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 (NCI-CTCAE v4.03) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies, with the exception of alopecia. The exceptions for such effects are allowed lab values of ≤Grade 2 specified elsewhere in these inclusion criteria.
* Life expectancy of at least 12 weeks.
* Able to swallow and retain oral medication.
* Participants must give informed consent according to the rules and regulations of the individual participating sites.
* Negative serum pregnancy test in women of childbearing potential within 14 days of first dose of treatment, and participants of childbearing potential must agree to use effective contraception during treatment up to 3 months from last dose. Fertile male partners must be willing and able to use effective non-hormonal means of contraception (barrier method of contraception in conjunction with spermicidal jelly, or surgical sterilization) during and for at least 6 months post-study treatment.
* The participant must be recovered from any prior treatment/major operation. The treatment/major operation must be performed at least 4 weeks prior to start of study drug. Palliative radiotherapy is permitted until one week prior to the start of study drug.
* Only incurable participants with histologically or cytologically proven primary tumor and objective documentation of disease progression on prior treatment by computerized tomography (CT)/ magnetic resonance imaging (MRI) may be enrolled.
* Ovarian, fallopian tube, or peritoneal carcinoma: both platinum refractory* and platinum resistant** participants, who have received ≥1 line of chemotherapy for relapsed disease (i.e., ≥2 lines of chemotherapy in total).

  *Platinum refractory is defined as progression during or within 4 weeks of last treatment with a platinum-containing therapy.

  **Platinum resistant is defined as relapse 4 weeks to <6 months after a platinum-containing therapy.
* Endometrial carcinoma: participants must have received ≥1 line of chemotherapy for relapsed or advanced (Stage IV, IIIc) disease.
* Cervical carcinoma: participants must have received ≥1 line of chemotherapy for relapsed or advanced (Stage IV b) disease.
* Carcinosarcomas (Malignant Mixed Mullerian Tumor) are allowed, but all other nonepithelial cancers of the ovary, fallopian tube, endometrium, or cervix are excluded.
* Participants must have either measurable disease per RECIST 1.1 or evaluable disease outside irradiated field on CT/MRI. For ovarian cancer: Participants must have disease that is measurable according to RECIST or assessable according to the Gynecological Cancer Intergroup (GCIG) CA-125 criterion. A rise in CA-125 or other tumor marker alone is not sufficient.

Exclusion Criteria:

* Disease-Specific Exclusions:

  * Evidence of complete or partial bowel obstruction.
  * Need of Total Parenteral Nutrition.
* Participants who are pregnant or breast feeding.
* Radiation (except planned or on-going palliative radiation to bone outside of the region of measurable disease) ≤3 weeks prior to Cycle 1 Day 1.
* Chemotherapy, endocrine therapy, immunotherapy or any other systemic anti-cancer therapy (including investigational anti-cancer therapy) ≤3 weeks prior to Cycle 1 Day 1.
* Diagnosis or recurrence of invasive cancer other than the present cancer within 3 years (except basal or squamous cell carcinoma of the skin that has been definitively treated).
* Unstable cardiovascular function:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (e.g. ventricular tachycardia on anti-arrhythmics are excluded and 1st degree atrioventricular (AV) block or asymptomatic left anterior fascicular block (LAFB)/ right bundle branch block (RBBB) will not be excluded), or
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) Class ≥3, or myocardial infarction (MI) within 3 months of Cycle 1 Day 1.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to the first dose. Active infection with concurrent treatment is acceptable only if the participant is clinically stable.
* Significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea.
* Concurrent therapy with approved or investigational anti-cancer therapeutics.
* Medical, psychological, or social conditions that may interfere with the participant's participation in the study or evaluation of the study results.
* Known brain metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and glucocorticoids.
* All non-epithelial cancers of the ovary, fallopian tube, peritoneum, endometrium or cervix as well as neuro-endocrine tumors are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 116 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven - Universitair Ziekenhuis Leuven, Leuven, Belgium
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev

REFERENCES:
- [Derived] Vergote IB, Lund B, Peen U, Umajuridze Z, Mau-Sorensen M, Kranich A, Van Nieuwenhuysen E, Haslund C, Nottrup T, Han SN, Concin N, Unger TJ, Chai Y, Au N, Rashal T, Joshi A, Crochiere M, Landesman Y, Shah J, Shacham S, Kauffman M, Mirza MR. Phase 2 study of the Exportin 1 inhibitor selinexor in patients with recurrent gynecological malignancies. Gynecol Oncol. 2020 Feb;156(2):308-314. doi: 10.1016/j.ygyno.2019.11.012. Epub 2019 Dec 9. PMID 31822399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 09-April-2014 and 29-Mar-2017.
Pre-assignment Details: A total of 116 participants were enrolled out of which 2 participants discontinued the study before the start of the treatment (1 participant due to death and 1 participant due to other reason). Total 114 participants started the study treatment.
Groups:
- Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIWmg/m^2: Participants with ovarian carcinoma who were platinum refractory or platinum resistant and had received at least one line of chemotherapy for relapsed disease received a dose of 35 mg/m^2 of selinexor oral tablets BIW (doses at least 36 hours apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 6 weeks of treatment, a dose of 50 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
Period: Overall Study
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIWmg/m^2 | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Started | 25 | 23 | 25 | 21 | 20
Modified Intent-to-treat(mITT)Population | 23 | 22 | 25 | 21 | 20
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 25 | 23 | 25 | 21 | 20
Not completed — Consent withdrawn | 0 | 0 | 1 | 0 | 0
Not completed — Termination of study by Sponsor | 4 | 3 | 1 | 1 | 3
Not completed — Death | 21 | 20 | 23 | 20 | 17

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on safety population that included all participants who had received any amount of study drug.
Groups:
- Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW: Participants with ovarian carcinoma who were platinum refractory or platinum resistant and had received at least one line of chemotherapy for relapsed disease received a dose of 50 mg/m^2 of selinexor oral tablets BIW (doses at least 36 hours apart) with light meal and 120 mL of water in a 4-week treatment cycles. After 12 weeks of treatment, a dose of 60 mg/m^2 of selinexor oral tablets BIW were administrated if the participants had no major toxicity. During dose reduction, participants received a minimum dose of 35 mg/m^2 QW. This treatment continued until PD or unacceptable toxicity or any discontinuation criteria or withdrawal of consent by the participant, or non-compliance by the participant with protocol requirements.
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW | Total
Number analyzed (Participants) | 25 | 23 | 25 | 21 | 20 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 6 | 20 | 13 | 14 | 70
  >=65 years | 8 | 17 | 5 | 8 | 6 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 25 | 21 | 20 | 114
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 23 | 25 | 21 | 20 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 25 | 23 | 24 | 21 | 20 | 113
  Race: Other-unspecified | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Control Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Disease Control Rate (DCR) was defined as the point estimate of the percentage of participants who had complete response (CR), partial response (PR), or stable disease (SD) for at least 12 weeks, assessed according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Participants without documented disease progression were censored on the date of last radiologic assessment.
Time Frame: Baseline up to 30 days after last dose administration, assessed after 6 weeks and 12 weeks (approximately 35 months)
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all participants who received at least 1 dose of study drug, had measurable disease per RECIST at baseline, and had at least 1 post-baseline efficacy follow-up information.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
percentage of participants | 30.4 [13.2 to 52.9] | 36.4 [17.2 to 59.3] | 24.0 [9.4 to 45.1] | 33.3 [14.6 to 57.0] | 30.0 [11.9 to 54.3]

2. Secondary Outcome: Percentage of Participants With Overall Response According to RECIST v1.1
Description: Overall Response Rate (ORR) was defined as the point estimate of the percentage of participants who had CR or PR, assessed according to RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline up to the date of progression or recurrence (approximately 35 months)
Population: Analysis was performed on mITT population that included all participants who received at least 1 dose of study drug, had measurable disease per RECIST at baseline, and had at least 1 post-baseline efficacy follow-up information.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
percentage of participants | 8.7 [1.1 to 28.0] | 13.6 [2.9 to 34.9] | 4.0 [0.1 to 20.4] | 9.5 [1.2 to 30.4] | 15.0 [3.2 to 37.9]

3. Secondary Outcome: Percentage of Participants With Disease Control According to Gynecological Cancer Intergroup (GCIG) Response Criteria
Description: DCR was defined as the point estimate of the percentage of participants who had CR, PR, or SD for at least 12 weeks, assessed according to GCIG response criteria (RECIST v1.1 and CA-125).
Time Frame: Baseline up to 30 days after last dose administration, assessed after 6 weeks and 12 weeks (approximately 35 months)
Population: Analysis was performed on GCIG evaluable population that included all participants in the ovarian cancer cohort (Cohort A) who had received at least 1 dose of study drug, had measurable disease per RECIST at baseline or baseline CA-125 assessment, and had at least 1 post-baseline efficacy follow-up information (i.e., either post-baseline scan or CA-125 assessment). Data for this outcome measure was not planned to be collected and analyzed for Cohort B and Cohort C, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 25 | 16 | 20
percentage of participants | 16.0 [4.5 to 36.1] | 23.8 [8.2 to 47.2] | 20.0 [5.7 to 43.7]

4. Secondary Outcome: Percentage of Participants With Overall Response According to GCIG Response Criteria
Description: ORR was defined as the point estimate of the percentage of participants who had CR or PR, assessed according to GCIG response criteria (RECIST v1.1 and CA-125).
Time Frame: Baseline up to the date of progression or recurrence (approximately 35 months)
Population: Analysis was performed on GCIG evaluable population that included all participants in the ovarian cancer cohort (Cohort A) who had received at least 1 dose of study drug, had measurable disease per RECIST at baseline or baseline CA-125 assessment, and had at least 1 post-baseline efficacy follow-up information (i.e., either post-baseline scan or CA-125 assessment). Data for this outcome measure were not planned to be collected and analyzed for Cohort B and Cohort C, as pre-specified in protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 25 | 21 | 20
percentage of participants | 4.0 [0.1 to 20.4] | 9.5 [1.2 to 30.4] | 10.0 [1.2 to 31.7]

5. Secondary Outcome: Progression-free Survival (PFS) According to RECIST v1.1
Description: PFS was defined as the time from date of start of study therapy to the date of tumor disease progression (i.e., radiological only) or date of death due to any cause. Participants without documented disease progression were censored at the time of last radiologic assessment. Participants without any post baseline assessments were censored at date of start of study therapy.
Time Frame: From start of study drug administration until PD or discontinuation from the study or death, whichever occurred first (approximately 35 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
days | 79.0 [45.0 to 99.0] | 86.5 [43.0 to 182.0] | 44.0 [43.0 to 141.0] | 85.0 [44.0 to 148.0] | 44.5 [43.0 to 140.0]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from the date of start of study therapy to the date of death due to any cause. Participants who were alive at the time of the analysis or were lost to follow-up were censored at the day they were last known to be alive. Kaplan-Maier method was used for estimation.
Time Frame: From start of study treatment up to the date of death, assessed every 3 months (approximately 35 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
days | 172.0 [62.0 to 372.0] | 226.0 [111.0 to 449.0] | 152.0 [83.0 to 254.0] | 348.0 [149.0 to 401.0] | 173.0 [105.0 to 353.0]

7. Secondary Outcome: Percentage of Participants Who Survived at 12 and 24 Months
Description: OS rate was reported as the percentage of participants who were alive at 12 and 24 months. OS was defined as time from the date of start of study therapy to the date of death due to any cause. Participants who were alive at the time of the analysis or are lost to follow-up were censored at the day they were last known to be alive. Survival rate were estimated by Kaplan-Maier method.
Time Frame: 12 and 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
percentage of participants
  12 months | 34.8 [16.6 to 53.7] | 31.8 [14.2 to 51.1] | 13.2 [3.4 to 29.9] | 33.3 [14.9 to 53.1] | 25.0 [9.1 to 44.9]
  24 months | 21.7 [7.9 to 39.9] | 13.6 [3.4 to 30.9] | 4.4 [0.3 to 18.4] | 19.0 [5.9 to 37.7] | 15.0 [3.7 to 33.5]

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE) and Treatment-emergent Serious Adverse Events (TESAE) According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not it is considered related to the medicinal product. A serious adverse event (SAE) was defined as an AE that meets one or more of the mentioned criteria, i.e., fatal, life threatening (places the participants at immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events. TEAE was defined as any AE (serious/non-serious) with onset or worsening of a pre-existing condition on or after the first administration of study medication through 30 days following last dose or any event considered drug-related by the investigator through the end of the study.
Time Frame: From start of study treatment up to 30 days after the last dose administration (approximately 35 months)
Population: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 25 | 23 | 25 | 21 | 20
Participants
  Participants with TEAE | 25 | 23 | 25 | 21 | 20
  Participants with TESAE | 14 | 14 | 6 | 12 | 12

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events by Severity According to National Cancer Institute Common Terminology Criteria for Adverse Events NCI CTCAE, Version 4.03
Description: AE: any unfavorable and unintended sign, symptom, or disease temporally associated with use of medicinal product, whether or not it is considered related to medicinal product. TEAE: any AE (serious/non-serious) with onset or worsening of a pre-existing condition on or after the first administration of study drug through 30 days following last dose or any event considered drug-related by investigator through end of study. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From start of study treatment up to 30 days after the last dose administration (approximately 35 months)
Population: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 25 | 23 | 25 | 21 | 20
Participants
  Mild (Grade 1) | 0 | 0 | 0 | 0 | 0
  Moderate (Grade 2) | 3 | 3 | 5 | 5 | 7
  Severe (Grade 3) | 19 | 17 | 17 | 15 | 13
  Life threatening (Grade 4) | 3 | 2 | 2 | 1 | 0
  Fatal (Grade 5) | 0 | 1 | 1 | 0 | 0

10. Secondary Outcome: Quality of Life (QoL): Change From Baseline European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQC30) Scores
Description: EORTC QLQC30: Disease specific indication that rates overall QoL in cancer participants. It consists of 30 general questions from 3 domains; 1) global health status, 2) functioning scales (physical, emotional, cognitive, social and role functioning), 3) symptom scales (fatigue, nausea, vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhea, financial difficulty). Out of 30 questions, 28 questions were scored using scale of 1 to 4, represented answers of 'not at all', 'a little', 'quite a bit', and 'very much'; remaining 2 questions contributed to global health status were scored on scale of 1 to 7, represented range of 'very poor' to 'excellent' that evaluated overall health and QoL. All scales and single-item measures range from 0 to 100, where higher score represented higher response level. Higher score for functional scale, global health status and symptom scale represented high level of functioning, high QoL, and high level of symptoms or problems, respectively.
Time Frame: Baseline, End of treatment (EOT) i.e., 30 days after last dose of study drug administration (up to 31 months)
Population: Analysis was performed on mITT population that included all participants who received at least 1 dose of study drug, had measurable disease per RECIST at baseline, and had at least 1 post-baseline efficacy follow-up information. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure and "Number analyzed' signifies number of participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 21 | 21 | 22 | 21 | 20
scores on a scale
  Global Health Status/ QoL: Baseline | 52.8 (22.41) | 59.5 (20.63) | 60.2 (24.25) | 61.5 (22.89) | 57.5 (21.95)
  Global Health Status/ QoL: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Global Health Status/ QoL: EOT | -8.3 (11.79) | -11.4 (29.88) | -14.6 (10.49) | -27.4 (31.81) | -13.9 (15.52)
  Functioning Scales/ Physical Functioning: Baseline | 69.5 (19.16) | 70.9 (21.54) | 66.1 (26.02) | 67.1 (21.14) | 70.7 (25.26)
  Functioning Scales/ Physical Functioning: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Functioning Scales/ Physical Functioning: EOT | -26.7 (28.28) | -16.4 (27.55) | -24.2 (21.32) | -7.6 (16.97) | -18.9 (14.25)
  Functioning Scales/ Role Functioning: Baseline: number analyzed (Participants) | 21 | 21 | 21 | 21 | 20
  Functioning Scales/ Role Functioning: Baseline | 54.0 (29.77) | 59.5 (31.87) | 55.6 (35.49) | 59.5 (28.66) | 63.3 (34.45)
  Functioning Scales/ Role Functioning: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Functioning Scales/ Role Functioning: EOT | -33.3 (47.14) | -3.0 (49.90) | -20.8 (36.96) | -9.5 (39.51) | -25.0 (9.13)
  Functioning Scales/ Emotional Functioning: Baseline | 62.3 (24.81) | 69.8 (24.65) | 71.2 (23.81) | 74.2 (19.53) | 66.3 (23.33)
  Functioning Scales/ Emotional Functioning: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Functioning Scales/ Emotional Functioning: EOT | -16.7 (11.79) | -0.8 (38.27) | 12.5 (14.43) | -13.9 (23.07) | -2.8 (17.21)
  Functioning Scales/ Cognitive Functioning: Baseline | 81.0 (22.54) | 86.5 (16.35) | 83.3 (25.20) | 83.3 (19.00) | 80.8 (23.12)
  Functioning Scales/ Cognitive Functioning: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Functioning Scales/ Cognitive Functioning: EOT | -33.3 (23.57) | -6.1 (29.13) | 4.2 (20.97) | -16.7 (38.49) | 0.0 (0.00)
  Functioning Scales/ Social Functioning: Baseline | 61.1 (29.97) | 76.2 (32.31) | 72.7 (28.89) | 69.0 (30.86) | 77.5 (29.75)
  Functioning Scales/ Social Functioning: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Functioning Scales/ Social Functioning: EOT | -33.3 (0.00) | -6.1 (48.46) | -20.8 (20.97) | -7.1 (18.90) | -30.6 (32.35)
  Symptom Scales/Items/ Fatigue: Baseline | 46.6 (27.80) | 43.4 (27.42) | 44.9 (27.75) | 46.0 (27.28) | 41.7 (27.89)
  Symptom Scales/Items/ Fatigue: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Fatigue: EOT | 33.3 (47.14) | 6.1 (41.09) | 1.4 (17.20) | 23.8 (30.38) | 16.7 (11.65)
  Symptom Scales/Items/ Nausea And Vomiting: Baseline | 13.5 (24.51) | 17.5 (30.04) | 9.8 (15.99) | 5.6 (14.27) | 10.8 (21.81)
  Symptom Scales/Items/ Nausea And Vomiting: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Nausea And Vomiting: EOT | 8.3 (11.79) | -0.0 (40.82) | 16.7 (19.25) | 9.5 (23.29) | 13.9 (16.39)
  Symptom Scales/Items/ Pain: Baseline | 34.9 (27.84) | 37.3 (27.34) | 32.6 (27.93) | 31.0 (29.48) | 32.5 (26.75)
  Symptom Scales/Items/ Pain: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Pain: EOT | -8.3 (11.79) | -4.5 (21.20) | 4.2 (8.33) | -2.4 (17.82) | 2.8 (26.70)
  Symptom Scales/Items/ Dyspnoea: Baseline: number analyzed (Participants) | 21 | 21 | 22 | 20 | 20
  Symptom Scales/Items/ Dyspnoea: Baseline | 23.8 (31.87) | 30.2 (36.37) | 19.7 (30.27) | 33.3 (38.01) | 21.7 (29.17)
  Symptom Scales/Items/ Dyspnoea: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Dyspnoea: EOT | 50.0 (23.57) | 6.1 (32.72) | 8.3 (16.67) | -0.0 (47.14) | 16.7 (18.26)
  Symptom Scales/Items/ Insomnia: Baseline | 31.7 (34.12) | 36.5 (31.46) | 30.3 (32.38) | 20.6 (26.82) | 38.3 (29.17)
  Symptom Scales/Items/ Insomnia: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Insomnia: EOT | -16.7 (23.57) | -9.1 (30.15) | -16.7 (33.33) | -19.0 (26.23) | 5.6 (32.77)
  Symptom Scales/Items/ Appetite Loss: Baseline | 25.4 (31.46) | 34.9 (32.45) | 30.3 (36.96) | 23.8 (28.17) | 15.0 (27.52)
  Symptom Scales/Items/ Appetite Loss: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Appetite Loss: EOT | 16.7 (23.57) | 0.0 (53.75) | 16.7 (43.03) | 33.3 (47.14) | 16.7 (34.96)
  Symptom Scales/Items/ Constipation: Baseline | 27.0 (27.12) | 15.9 (24.99) | 15.2 (26.68) | 17.5 (30.95) | 11.7 (16.31)
  Symptom Scales/Items/ Constipation: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Constipation: EOT | 0.0 (47.14) | 6.7 (43.89) | 8.3 (16.67) | 9.5 (31.71) | -5.6 (13.61)
  Symptom Scales/Items/ Diarrhoea: Baseline | 17.5 (30.95) | 9.5 (26.13) | 18.2 (24.62) | 18.3 (31.48) | 8.3 (14.81)
  Symptom Scales/Items/ Diarrhoea: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Diarrhoea: EOT | 0.0 (0.00) | -3.0 (34.82) | 0.0 (27.22) | 23.8 (25.20) | 27.8 (32.77)
  Symptom Scales/Items/ Financial Difficulties: Baseline | 7.9 (17.97) | 4.8 (15.94) | 16.7 (26.73) | 9.5 (18.69) | 5.0 (12.21)
  Symptom Scales/Items/ Financial Difficulties: EOT: number analyzed (Participants) | 2 | 11 | 4 | 7 | 6
  Symptom Scales/Items/ Financial Difficulties: EOT | 16.7 (23.57) | 3.0 (17.98) | 0.0 (0.00) | 4.8 (29.99) | -5.6 (13.61)

11. Secondary Outcome: Number of Participants With Individual Clinically Significant Abnormalities in Laboratory Tests
Description: Clinically significant laboratory tests abnormalities were analyzed and reported for this outcome measure.
Time Frame: From start of study treatment up to 30 days after the last dose administration (approximately 35 months)
Population: Analysis was performed on safety population that included all participants who had received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
Number analyzed (Participants) | 23 | 22 | 25 | 21 | 20
Participants | 21 | 20 | 19 | 14 | 11

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after last dose administration (approximately 35 months)
Description: Analysis was performed on safety population that included all participants who had received any amount of study medication.
Arm/Group | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW
All-Cause Mortality (participants affected / at risk) | 21/25 | 20/23 | 23/25 | 20/21 | 17/20
Serious Adverse Events (participants affected / at risk) | 14/25 | 14/23 | 6/25 | 12/21 | 12/20
Other Adverse Events (participants affected / at risk) | 25/25 | 23/23 | 25/25 | 21/21 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=25) | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=23) | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=25) | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW (N=21) | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW (N=20)
Vomiting (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 4
Ileus (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Varicella Zoster Virus Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Escherichia Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 0 | 0 | 0 | 2
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Drain Placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Cohort A-Ovarian Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=25) | Part 1: Cohort B-Endometrial Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=23) | Part 1: Cohort C-Cervical Carcinoma: Selinexor up to 60 mg/m^2 BIW (N=25) | Part 2: Cohort A-Ovarian Carcinoma Schedule 1: Selinexor up to 50 mg/m^2 BIW (N=21) | Part 2: Cohort A-Ovarian Carcinoma Schedule 2: Selinexor up to 60 mg/m^2 QW (N=20)
Nausea (Gastrointestinal disorders) | 22 | 15 | 17 | 17 | 15
Vomiting (Gastrointestinal disorders) | 18 | 14 | 11 | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 6 | 10 | 8
Abdominal Pain (Gastrointestinal disorders) | 7 | 1 | 3 | 5 | 7
Abdominal Distension (Gastrointestinal disorders) | 3 | 1 | 2 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 1 | 3 | 1
Ascites (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 5
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Defaecation Urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal Irritation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral Mucosal Blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 12 | 15 | 15 | 14 | 14
Asthenia (General disorders) | 7 | 7 | 5 | 6 | 3
Malaise (General disorders) | 3 | 3 | 2 | 1 | 2
Pyrexia (General disorders) | 3 | 1 | 4 | 3 | 1
Oedema Peripheral (General disorders) | 3 | 2 | 2 | 6 | 2
Face Oedema (General disorders) | 2 | 2 | 2 | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 2 | 0 | 1 | 1
Oedema (General disorders) | 2 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 12 | 18 | 12 | 16 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 8 | 3 | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5 | 3 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5 | 2 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 0 | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 13 | 11 | 14 | 9 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 10 | 13 | 4 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 7 | 5 | 11 | 4 | 6
Dizziness (Nervous system disorders) | 7 | 5 | 6 | 4 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 4 | 3 | 0 | 3
Headache (Nervous system disorders) | 3 | 1 | 3 | 1 | 4
Paraesthesia (Nervous system disorders) | 0 | 2 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 12 | 13 | 18 | 11 | 6
Urinary Tract Infection (Infections and infestations) | 4 | 2 | 2 | 2 | 2
Cystitis (Infections and infestations) | 2 | 3 | 1 | 1 | 1
Lung Infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes Simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 7 | 8 | 5 | 7 | 5
Visual Impairment (Eye disorders) | 2 | 1 | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6 | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 3 | 5
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 7 | 1 | 5 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 3 | 2 | 0
Confusional State (Psychiatric disorders) | 1 | 2 | 2 | 2 | 1
Depression (Psychiatric disorders) | 1 | 1 | 2 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 4 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 3 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 4 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 2 | 2 | 0 | 3 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 2 | 3 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 1 | 3 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 0 | 2 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 1 | 1
Auditory Disorder (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 2 | 1 | 1
Device Occlusion (Product Issues) | 2 | 0 | 2 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 7 | 6 | 6 | 11 | 7
Device Related Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Polyurea (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT02025985/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT02025985/SAP_001.pdf